CLINICAL TRIAL: NCT02203500
Title: Tolerability and Pharmacokinetics of 80 mg Telmisartan and 6 mg Lacidipine Alone and in Combination After 7 Days Treatment. An Open Randomised Three-way Cross-over Trial in Female and Male Healthy Subjects
Brief Title: Tolerability and Pharmacokinetics of Lacidipine With and Without the Co-administration of Telmisartan in Female and Male Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1173.2
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — lacidipine; Telmisartan

ARMS (3):
- Lacidipine (Experimental)
  Interventions: Drug: Lacidipine
- Telmisartan (Experimental)
  Interventions: Drug: Telmisartan
- Lacidipine + Telmisartan (Experimental)
  Interventions: Drug: Lacidipine; Drug: Telmisartan

INTERVENTIONS:
Drug: Lacidipine
  Arms: Lacidipine; Lacidipine + Telmisartan
Drug: Telmisartan
  Arms: Lacidipine + Telmisartan; Telmisartan

SUMMARY:
The objectives of this study are to compare the steady state pharmacokinetics of lacidipine with and without the co-administration of telmisartan and to compare the steady state pharmacokinetics of telmisartan with and without the co-administration of lacidipine

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female Caucasian subjects as determined by results of screening
* Written informed consent in accordance with Good Clinical Practice and local legislation given
* Age >= 18 and <= 50 years
* Broca >= -20% and <= + 20%

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and Electrocardiogram (ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurologic disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (<= 1 month prior to administration or during the trial)
* Use of any drugs which might influence the results of the trial (<= 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (<= 2 months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 60g/day)
* Drug abuse
* Blood donation > 100 ml (<= 4 weeks prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance
* Female only:

  * no reliable contraception (reliable are: oral contraceptives, 3-month injection, Intrauterine devices (IUD), sterilization)
  * Pregnancy or breast feeding period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 1998-10; Primary Completion 1999-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects with clinically significant changes in vital signs | up to 12 days after last drug administration
Number of subjects with abnormal changes in laboratory parameters | up to 12 days after last drug administration
Cmax (Maximum measured concentration of the analyte in plasma) | up to 72 hours after drug administration
Cmin (Minimum measured concentration of the analyte in plasma) | up to 72 hours after drug administration
AUCss (Area under the concentration-time curve of the analyte in plasma at steady state) | up to 72 hours after drug administration
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 72 hours after drug administration
CL/F (Apparent clearance of the analyte in plasma following extravascular administration) ) | up to 72 hours after drug administration
Vz/F (Apparent volume of distribution of the analyte during the terminal phase) | up to 72 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 72 hours after drug administration
MRT (Mean residence time of the analyte in the body) | up to 72 hours after drug administration
Number of subjects with adverse events | up to 66 days